CLINICAL TRIAL: NCT04206020
Title: A Phase 3, Multi-Center, Randomized, Double-Masked, Placebo-Controlled Study of Safety and Efficacy of SkQ1 Ophthalmic Solution in the Environment and the Controlled Adverse Environmental (CAE®) Model for the Treatment of Dry Eye Syndrome
Brief Title: Vehicle-Controlled Study of SkQ1 as Treatment for Dry-eye Syndrome
Acronym: VISTA-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mitotech, SA (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-110-0011
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Results first posted 2022-01-19 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-12

CONDITIONS: Dry Eye Syndrome
Keywords: Dry Eye; Dry Eye Syndrome; SkQ1; KCS; Keratoconjunctivitis
MeSH Terms: conditions — Dry Eye Syndromes; Keratoconjunctivitis | interventions — Visomitin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Parallel-group study SkQ1 Ophthalmic Solution versus placebo (vehicle) solution
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator: SkQ1 Vehicle (Placebo Comparator): Vehicle for SkQ1 Ophthalmic Solution
  Interventions: Drug: SkQ1 Vehicle Solution
- SkQ1 (Active Comparator): SkQ1 Ophthalmic Solution
  Interventions: Drug: SkQ1 Ophthalmic Solution

INTERVENTIONS:
Drug: SkQ1 Vehicle Solution — SkQ1 Ophthalmic Solution Vehicle
  Other Names: Vehicle for SkQ1
  Arms: Placebo Comparator: SkQ1 Vehicle
Drug: SkQ1 Ophthalmic Solution — SkQ1 Ophthalmic Solution
  Other Names: Visomitin
  Arms: SkQ1

SUMMARY:
The purpose of this study is to evaluate whether SkQ1 Ophthalmic Solution is safe and effective compared to Vehicle for the treatment of the signs and symptoms of dry eye syndrome.

DETAILED DESCRIPTION:
Multi-center, double-masked, randomized, placebo-controlled study comprising 5 visits over the course of approximately 9 weeks. Qualified subjects are randomized 1:1 to receive either SkQ1 Ophthalmic Solution, or Placebo (vehicle of SkQ1 Ophthalmic Solution).

The Primary Endpoints are:

Change from Baseline (Visit 2) to Visit 5 of Ocular Discomfort;

Change from Baseline (Visit 2) to Visit 5 of conjunctival fluorescein staining (sum of temporal and nasal regions)

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age;
* Provide written informed consent;
* Have a subject reported history of dry eye;
* Have a history of use of eye drops for dry eye symptoms;
* Ocular Discomfort;
* Schirmer's Test score;
* Have corneal fluorescein staining ;
* Have lissamine green conjunctival Staining;
* Have a conjunctival redness;

Exclusion Criteria:

* Have been previously exposed to previous SkQ1 Ophthalmic Solution treatment;
* Have any clinically significant slit lamp findings at Visit 1;
* Be diagnosed with an ongoing ocular infection or active ocular inflammation at Visit 1;
* Have had any ocular and/or lid surgeries within 6 months of Visit 1 or any planned over the study period;
* Have an uncontrolled systemic disease;
* Be a woman who is pregnant, nursing or planning a pregnancy;
* Be a woman of childbearing potential who is not using an acceptable means of birth control;
* Have a known allergy and/or sensitivity to the study drug or its components;
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation
Enrollment: 610 (Actual)
Dates: Start 2019-12-20 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence T Friedhoff, MD, PhD, Study Chair — Mitotech, SA
Locations (4):
- United States (4):
  - Arizona Eye Institute and Cosmetic Laser, Sun City West, Arizona
  - Andover Eye Associates, Andover, Massachusetts
  - Eye Clinics of South Texas, San Antonio, Texas
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SkQ1 Ophthalmic Solution: SkQ1 Ophthalmic Solution (1.55µg/mL)
Period: Overall Study
Arm/Group | Placebo Comparator: SkQ1 Vehicle | SkQ1 Ophthalmic Solution
Started | 306 | 304
Completed | 298 | 297
Not Completed | 8 | 7
Not completed — Adverse Event | 1 | 4
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Pregnancy | 0 | 1
Not completed — Unable to attend visits | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Comparator: SkQ1 Vehicle | SkQ1 Ophthalmic Solution | Total
Number analyzed (Participants) | 306 | 304 | 610
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 166 | 150 | 316
  >=65 years | 140 | 154 | 294
Age, Continuous [Mean (Standard Deviation); unit: years]
  Mean (SD) | 61.9 (11.92) | 62.8 (12.58) | 62.4 (12.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 209 | 432
  Male | 83 | 95 | 178
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 13 | 11 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 50 | 34 | 84
  White | 241 | 253 | 494
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 306 | 304 | 610
Ocular Discomfort Scale [Mean (Standard Deviation); unit: units on a scale] | 2.7 (1.06) | 2.7 (0.98) | 2.7 (1.02)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Discomfort Scale
Description: Change of Ocular Discomfort Scale, scale ranged from 0 to 4 with 0 = No Discomfort and 4 = Constant Discomfort.
Time Frame: From baseline to Day 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Comparator: SkQ1 Vehicle | SkQ1 Ophthalmic Solution
Number analyzed (Participants) | 306 | 304
units on a scale | -0.6 (1.36) | -0.6 (1.34)

2. Primary Outcome: Conjunctival Fluorescein Staining
Description: Change of Conjunctival Fluorescein Staining (sum of temporal and nasal regions), scale in each region ranged from 0 to 4 with 0 = No Staining and 4 = Confluent Staining
Time Frame: From baseline to Day 57
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Comparator: SkQ1 Vehicle | SkQ1 Ophthalmic Solution
Number analyzed (Participants) | 251 | 250
units on a scale | -0.63 (1.087) | -0.69 (1.150)

ADVERSE EVENTS:
Time Frame: From Day -7 through end of study (Day 57)
Arm/Group | Placebo Comparator: SkQ1 Vehicle | SkQ1 Ophthalmic Solution
All-Cause Mortality (participants affected / at risk) | 0/306 | 0/304
Serious Adverse Events (participants affected / at risk) | 2/306 | 2/304
Other Adverse Events (participants affected / at risk) | 19/306 | 20/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator: SkQ1 Vehicle (N=306) | SkQ1 Ophthalmic Solution (N=304)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Comparator: SkQ1 Vehicle (N=306) | SkQ1 Ophthalmic Solution (N=304)
Instillation site pain (General disorders) | 13 (18) | 15 (19)
Visual acuity reduced (Eye disorders) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Authorship and manuscript composition will reflect cooperation among all parties involved in the study. Authorship will be established before writing the manuscript. The study sponsor will have the final decision regarding the manuscript and publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/20/NCT04206020/Prot_SAP_000.pdf